CLINICAL TRIAL: NCT02219828
Title: AnakInRa for Treatment of Recurrent Idiopathic Pericarditis
Brief Title: AnakInRa for Treatment of Recurrent Idiopathic Pericarditis (AIRTRIP)
Acronym: AIR TRIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massimo Imazio (Other)
Responsible Party: Sponsor-Investigator, Massimo Imazio, Cardiology Dpt ASLTO2, Maria Vittoria Hospital
Organization: Maria Vittoria Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 40/08/13; 2013-001849-13 (EudraCT Number)
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Idiopathic Recurrent Pericarditis
Keywords: pericarditis; recurrent pericarditis; corticosteroids; anakinra
MeSH Terms: conditions — Pericarditis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo sc
  Interventions: Drug: Placebo
- Anakinra (Active Comparator): Anakinra 2mg/Kg up to 100mg (maximum dose)
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — 2mg/Kg daily sc up to 100mgday as maximum dose
  Arms: Anakinra
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Recent findings suggest that recurrent pericarditis (RP) may be a previously unrecognized autoinflammatory disease. The pivotal pathogenic role of interleukin (IL)-1 in RP has been shown by the achievement of complete responses after treatment with the recombinant IL-1-receptor antagonist, anakinra. Anakinra is the recombinant form of IL-1Ra. The proposed study is designed to demonstarate the efficacy of anakinra in RP.

DETAILED DESCRIPTION:
This is a 8-month, multicenter (3 Italian centers), randomized, double-blind, placebo-controlled, multicenter, medication-withdrawal study to evaluate the efficacy, tolerability, and safety of anakinra in adults and children with idiopathic recurrent pericarditis (RP).

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written informed consent for ≥ 18 years of age before any assessment is performed. Parents' or legal guardian's written informed consent and child's assent, if appropriate, are required before any assessment is performed for patients < 18 years of age.
2. Age > 2 years and <70 years at screening visit;
3. Recurrent pericarditis defined as a first episode of acute pericarditis followed by recurrences (Ann Intern Med. 2011;155:409-14) (at least two recurrences for this study). First episode of pericarditis is diagnosed when at least two of the following criteria were present: pericarditic typical chest pain (sharp and pleuritic, improved by sitting up and leaning forward), pericardial friction rubs, widespread ST segment elevation or PR depressions not previously reported, and new or worsening pericardial effusion. Recurrence is diagnosed when chest pain recurs and one or more of the following signs is present: fever, pericardial friction rub, ECG changes, echocardiographic evidence of new or worsening pericardial effusion, and elevations in the white blood cell count, erythrocyte sedimentation rate or C-reactive protein. To be enrolled in this study, elevation of C-reactive protein is mandatory both in the first attack and in the following recurrences. We differentiate recurrences from incessant pericarditis, term used to define patients with continued activity of pericarditis (with a symptom-free interval of < 6 weeks) (Soler-Soler J, Sagristà-Sauleda J, Permanyer-Miralda G. Relapsing pericarditis. Heart. 2004;90:1364-8).
4. Specific etiologies excluded, including tuberculous, neoplastic or purulent etiologies, post-cardiac injury syndromes, and rheumatic autoimmune diseases.
5. Records to document the number of prior pericardial recurrences, the time interval between them as well as prior treatments must be made available from the medical charts.
6. Troponin values during at least one previous attack is recorded.
7. QuantiFERON (QFT-TB G In-Tube) test or positive Purified Protein Derivative (PPD) test has been previously made and recorded.
8. Patients will be enrolled at the time of a recurrent episode (at least the second recurrence, i.e. third episode) or "relapse" of pericarditis documented by the following criteria:

   * recurrent pericardial pain (with a score of least 5 on the 21 circles VAS) AND
   * increase in CRP≥1 mg/dL (being normal value = 0 - 0.5 mg/dL ), AND
   * one or more of the following signs: fever (≥ 37°C), pericardial friction rub, pertinent ECG changes, echocardiographic evidence of of new or worsening pericardial effusion (see definition above)
9. Continuous treatment with CS, the dose of which must not have been increased in the three days preceding enrolment
10. Women of child bearing potentials (WCBP), defined as pre-menarche females aged 8 years and above or all women physiologically capable of becoming pregnant, sexually active, must use an effective form of contraception. Medically approved contraception (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices) could include total abstinence. Reliable contraception should be maintained throughout the study and for 3 months after anakinra discontinuation. Women are considered post-menopausal and not WCBP if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. appropriate age, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks prior to study entry. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment she considered a WCBP.

Exclusion Criteria:

* Patients fulfilling any of the following criteria are not eligible for enrollment in this study:

  1. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
  2. History of being immunocompromised, including a positive HIV at screening (ELISA and Western blot) test result.
  3. Positive QuantiFERON (QFT-TB G In-Tube) test or positive Purified Protein Derivative (PPD) test (≥ 5 mm induration) performed after the first attack of pericarditis. Patients with a positive PPD test (≥ 5 mm induration) at screening may be enrolled only if they have either a negative chest X-ray or a negative QuantiFERON test.
  4. Live vaccinations within three months prior to the start of the trial, during the trial, and up to three months following the last anakinra dose.
  5. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
  6. History of significant other medical conditions, which in the Investigator's opinion would exclude the patient from participating in this trial including current pericarditis due to known diseases (e.g. tuberculosis, neoplastic or purulent causes, connective tissue diseases, acute rheumatic fever, etc.)
  7. History of recurrent and/or evidence of active bacterial, fungal, or viral infection(s).
  8. History of Type I hypersensitivity to anakinra.
  9. History of poor compliance.
  10. Use of any investigational drug (or biologic), or device within five half-lives of the drug prior to study entry or during the study.

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | 8 months
  Time to flare in the anakinra and placebo arms

SECONDARY OUTCOMES:
1. responder status in the open label phase | 60 days
  To assess the responder status in the open label phase at Day 8 and 60 and at the end of the study with the following three criteria all to be met:
  1. no or mild pericardial pain (a score ≤2.5 on a 21 circle VAS), AND
  2. normal CRP levels (CRP ≤0.5 mg/dL), AND
  3. absent or mild (≤10 mm) echocardiographic effusion. Assessments will be performed at Days 4, and 8 (study Period 1), and then at Day 30, and Months 2, 4, 6, and 8 if not otherwise specified.
2. change over time of the 3 outcome criteria, i.e. pericardial pain, CRP levels, and echocardiographic effusion; | 8 months
  Assessments will be performed at Days 4, and 8 (study Period 1), and then at Day 30, and Months 2, 4, 6, and 8 if not otherwise specified.
3. time to response in the open label phase | 8 months
  Assessments will be performed at Days 4, and 8 (study Period 1), and then at Day 30, and Months 2, 4, 6, and 8 if not otherwise specified.
4. percentage of patients who relapse in the withdrawal part in the two arms; | 8 months
  Assessments will be performed at Days 4, and 8 (study Period 1), and then at Day 30, and Months 2, 4, 6, and 8 if not otherwise specified.
5. change over time in patient's/parent's global assessment of overall well being on a 21 circle VAS; | 8 months
  Assessments will be performed at Days 4, and 8 (study Period 1), and then at Day 30, and Months 2, 4, 6, and 8 if not otherwise specified.
6. change over time in the global evaluation of disease activity by physicians on a 21 circle VAS | 8 months
  Assessments will be performed at Days 4, and 8 (study Period 1), and then at Day 30, and Months 2, 4, 6, and 8 if not otherwise specified.
8. percentage off CS and any other concurrent medication at 6weeks | 6 weeks
  Assessments will be performed at Days 4, and 8 (study Period 1), and then at Day 30, and Months 2, 4, 6, and 8 if not otherwise specified.
9. tolerability and safety of the treatment | 8 months
  To assess the tolerability and safety of the treatment, i.e. monitoring and recording all adverse events (AEs), with attention to local tolerability to s.c. injection, and serious adverse events (SAEs), and the regularly scheduled monitoring of hematology, blood chemistry, physical examinations, and vital signs including blood pressure over 8 months. Assessments will be performed at Days 4, and 8 (study Period 1), and then at Day 30, and Months 2, 4, 6, and 8 if not otherwise specified.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Internal Medicine Division, OSpedale Papa Giovanni XXIII, Bergamo, Bergamo
  - Pediatric Dept. Ospedale Gaslini, Genova, Genova
  - Cardiology Dpt, Maria Vittoria Hospital, Torino, Torino

REFERENCES:
- [Derived] Brucato A, Imazio M, Gattorno M, Lazaros G, Maestroni S, Carraro M, Finetti M, Cumetti D, Carobbio A, Ruperto N, Marcolongo R, Lorini M, Rimini A, Valenti A, Erre GL, Sormani MP, Belli R, Gaita F, Martini A. Effect of Anakinra on Recurrent Pericarditis Among Patients With Colchicine Resistance and Corticosteroid Dependence: The AIRTRIP Randomized Clinical Trial. JAMA. 2016 Nov 8;316(18):1906-1912. doi: 10.1001/jama.2016.15826. PMID 27825009